CLINICAL TRIAL: NCT01870479
Title: Music & Cancer - Live Music During Chemotherapy. Randomized Study of the Effect of Live Music During Chemotherapy Treatment
Brief Title: Music & Cancer - Live Music During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Margrethe Langer Bro (Other)
Collaborators: Danish Cancer Society (Other); University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Margrethe Langer Bro, Assistant professor, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-20120118
Record Dates: First submitted 2013-04-09; First posted 2013-06-06 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Non Hodgkin´s Lymphomas; Hodgkin´s Lymphomas
Keywords: Malignant Lymphoma; Chemotherapy; Music therapy
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Live music (Experimental): Patient preferred live music during chemotherapy session.
  Interventions: Other: Live music
- Taped music (Active Comparator): Patient preferred taped music during chemotherapy
  Interventions: Other: Taped music
- Control (No Intervention): Usual care during chemotherapy

INTERVENTIONS:
Other: Live music
  Arms: Live music
Other: Taped music
  Arms: Taped music

SUMMARY:
Main purpose: To determine if live music moderates the level of chemotherapy related anxiety, in patients with haematological cancer

The investigators hypothesize that live music:

1. Have an ameliorating effect on physical and psychological symptoms during chemotherapy treatment
2. May counteract the patients feeling of loss of identity and alienation in this particular group of cancer patients.
3. Is more effective in patients with good musical abilities.
4. Is more effective than taped music.

Method: Intervention groups:

1. Listening to patient-preferred live music during chemotherapy
2. Listening to patient-preferred taped music during chemotherapy
3. Standard care

Endpoints:

Primary: Level of anxiety measured by STAI. Secondary: Serum catecholamines.

Background: In order to establish the intervention procedures, the investigators have carried out a pilot study at the hematology department at Hospital of Southwest Denmark, including students from the Academy of Music and Dramatic Arts, Southern Denmark. The pilot results indicates that live music has an uplifting, pain relieving, and then releasing effect and that music has a positive impact on hospitalisation. According to the evaluation forms filled out by 243 cancer patients, the music experience has provided human anchorage/cohesion as a counterweight to disease fixation and alienation Chemotherapy involves major physical and psychological problems. Not much has been provided in the clinical setting which relieves the symptoms of anxiety associated with chemotherapy. A review of the literature illustrate the need for developing new potential areas of intervention that takes into account, that not only do cancer patients face challenges in everyday life ranging from physiological changes over social to psychological problems, but also during treatment procedures, which may cause a higher level of anxiety associated with these procedures, e.g., chemotherapy infusion.This project investigates to what degree live music may relieve some of these symptoms during treatment for haematological cancer. The project is created in order to both measure psychosocial effects as well as direct stress measures, i.e. serum catecholamine. These physiological changes are measured in order to shed light on the mechanism behind the potential effects of live music on discomfort in connection with chemotherapy treatment.

Perspectives: The vision of the project focus on strengthening the cancer patients' ability to cope with physiological and psychological issues during chemotherapy sessions and to make the patients conscious of music as an option in these coping efforts. Hopefully, the results will provide a scientific basis for an evaluation of the perspectives and the potentials of live music treatment during chemotherapy infusion among cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Newly diagnosed with malignant lymphoma and planned first line chemotherapy treatment
* Able to give informed consent

Exclusion Criteria:

* Patients who do not speak or understand Danish
* Patients who are deaf or blind.
* Any comorbidity that postpone planed chemotherapy for more than 4 weeks
* Patients with alcohol or drugs misuse problems as stated in the medical record.
* Patients with untreated mental illness as identified in the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Anxiety (STAI) | Measurement of STAI after the 5. chemotherapy (on average 8 weeks after inclusion)
  STAI-S Spielberger State-Trait Anxiety Scale-State

SECONDARY OUTCOMES:
Serum catecholamines | Measured before and after each chemotherapy (at baseline and on average after 2, 4, 6, and 8 weeks after inclusion)
  Blood samples
Nausea | Between each visit (at baseline and on average after 1, 3, 5, and 7 weeks after inclusion)
  Patient diary
Quality of life | Visit 1, 2, 4, 6, 7. (at basline and on average after 2, 4, 6, and 8 weeks after inclusion)
  Quality of Life Questionnaire: QLQ-C30
Anxiety (HADS) | Visit 1, 2, 3 and 4 (at baseline and on average 2, 4, 6 weeks after inclusion)
  Hospital Anxiety and Depression Scale (HADS)
Distress | Visit 1, 2, 4 and 6 (at basline and on average after 2, 4, 6, and 8 weeks after inclusion)
  questionaire: The Distress Thermometer
Anxiety (STAI) | Measurement of STAI at baseline and after each chemotherapy 1 to 5 (on average 2, 4, 6 and 8 weeks after inclusion) as well as differences from baseline.
  STAI-S Spielberger State-Trait Anxiety Scale-State

CONTACTS AND LOCATIONS:
Overall Officials: Margrethe L Bro, PhD student, Principal Investigator — IRS, Southern Denmark. Assistant professor at The Academy of Music in Southern Denmark
Locations (7):
- Denmark (7):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Hospital of Southwest Jutland, Esbjerg, Region of Southwest Denmark
  - Odense University Hospital, Odense, Region of Southwest Denmark
  - The Academy of Music and Dramatic Arts, Southern Denmark, Odense, Region of Southwest Denmark
  - Roskilde Sygehus, Roskilde, Region Sjælland
  - Rigshospitalet, Copenhagen, The Capital Region of Denmark
  - Herlev Hospital, Copenhagen, The Capital Region of Denmark